CLINICAL TRIAL: NCT04988841
Title: Prospective randomIzed Clinical Trial Assessing the Tolerance and Clinical Benefit of feCAl tranSplantation in patientS With melanOma Treated With CTLA-4 and PD1 Inhibitors
Brief Title: Assessing the Tolerance and Clinical Benefit of feCAl tranSplantation in patientS With melanOma
Acronym: PICASSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200133
Record Dates: First submitted 2021-06-25; First posted 2021-08-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
Keywords: Fecal microbiome transfer; Microbiome restoration biotherapeutic; Full-ecosystem intestinal microbiome; Response to anti- CTLA-4 and anti PD1; the tumor microenvironment; Peripheral blood T cell subpopulations; Efficacy and safety of MaaT013
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab; MoviPrep; Normacol

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized, double blinded, pilot, proof-of concept, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At week 27, unblinding will be performed on patients who progressed. For those who received Placebo, Maat 013 will be administrated in open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiotherapy (MaaT013) associated to ipilimumab and nivolumab (Experimental): Fecal microbiotherapy MaaT013 (actif arm) enemas will be administered by nurses, at the hospital, in the dermatology department in which the patients are treated for their melanoma. Nurses will be trained to administer enemas. The enema will be administered to the patient in the left lateral position with instructions to retain it for at least 20 minutes
  Interventions: Drug: MaaT013; Drug: Ipilimumab; Drug: Nivolumab; Drug: MoviPrep; Drug: Normacol
- fecal microbiotherapy Placebo associated to ipilimumab and nivolumab (Placebo Comparator): Placebo fecal microbiotherapy will be administered by nurses, at the hospital, in the dermatology department in which the patients are treated for their melanoma. Nurses will be trained to administer enemas. The enema will be administered to the patient in the left lateral position with instructions to retain it for at least 20 minutes
  Interventions: Drug: MaaT013; Drug: Ipilimumab; Drug: Nivolumab; Drug: MoviPrep; Drug: Normacol; Drug: Placebo of Maat013

INTERVENTIONS:
Drug: MaaT013 — study is an experimental drug , produced by MaaT Pharma, and composed of pooled-donor, full-ecosystem intestinal microbiome (455 species approximately against 274 on average)
  Other Names: fecal microbiotherapy
Drug: Ipilimumab — Anti cytotoxicT-lymphocyte-associated protein 4 ( immunothérapy)
Drug: Nivolumab — AntiPD1 ( immunothérapy)
Drug: MoviPrep — Osmotic laxative solution : patients take a single dose of two liters of Moviprep® or equivalent the night before the first administration of experimental treatment (Fecal microbiota transfer or placebo)
  Other Names: Osmotic laxative solution
Drug: Normacol — hypertonic enema solution
  Other Names: hypertonic enema solution
Drug: Placebo of Maat013 — expérimental drug placebo of MaaT013
  Other Names: fecal microbiotherapy placebo
  Arms: fecal microbiotherapy Placebo associated to ipilimumab and nivolumab

SUMMARY:
Recent studies suggest that patients with metastatic melanoma whose gut microbiome is colonized by eubiotic bacteria have a stronger anti-cancer response to anti CTLA-4 and anti PD1. The hypothesis of this research is that a pooled standardized fecal microbiome transfer (FMT) will shift melanoma patients' gut microbiome towards a composition close to that associated with a better response, and will therefore increase the response to a combination of anti CTLA-4 and anti PD1, without affecting the safety of these drugs. The present trial is the first randomized trial of FMT in patients with unresectable or metastatic melanoma. It will include patients who have neither been exposed to anti CTLA-4 nor anti PD1 or PDL-1, prior to inclusion in the study. The pooled standardized fecal microbiome transfer administered in this study is an experimental drug MaaT013, a microbiome restoration biotherapeutic, produced by MaaT Pharma, and composed of pooled-donor, full-ecosystem intestinal microbiome. The MaaT013 product has a standardized richness (in number of species present) higher than a product obtained from a mono donor (455 species approximately against 274 on average) and contains bacteria species (mentioned in the rationale) associated with better response to anti- CTLA-4 and anti PD1.

DETAILED DESCRIPTION:
PICASSO is a prospective, randomized, proof of concept clinical trial. This trial is about assessing the tolerance and clinical benefit of fecal microbiome transfer in patients with melanoma in addition to the usual treatment with immunotherapy combining ipilimumab (CTLA-4 inhibitor) and nivolumab (PD-1 inhibitor).

In the proposed research, we will compare faecal transplantation using MaaT013 to placebo in 70 patients.

Patients not exposed to anti CTLA-4 and anti PD1 or PDL-1 patients before the trial will be randomized to receive either: ipilimumab + nivolumab + MaaT013 (n = 35) or ipilimumab + nivolumab + placebo (n = 35).

The estimated duration of the study is 37 months. Administration of MaaT013 or placebo will be performed every 3 weeks between baseline and week 9 then from week 15 to week 23 every 4 weeks. A total of 7 fecal microbiome transfer will be performed.

Prior to the first administration (the day before) an evacuating enema by (MOVIPREP or equivalent) will be done, For subsequent administrations, an evacuating enema (equivalent to the specialty Normacol®) will be administered rectally before the transplantation of fecal microbiota or the placebo.

Blood and stool samples will be collected as well as biopsies for the purposes of the study.

An evaluation of the patient's condition will be made at week 27, Unblinding will be performed for patients who have progressed. Patients with disease progression who received placebo will be considered for receiving MaaT013, in an open-label basis, concurrently with nivolumab infusions, at week 31, 35, 39, 43 and 47.

. The end-of-follow-up visit for all patients is scheduled for week 51. Patients who met the inclusion criteria, received Ipilimumab+Nivolumab, who consented to have a baseline stool microbiota analysis before starting treatment with ipilimumab + nivolumab. They will form a cohort of 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80
* Patients with unresectable or metastatic melanoma
* Patients with ECOG performance of 0-2
* Patients able to provide written informed consent and understand the risks associated with MaaT013
* Have measurable disease as per RECIST version 1.1, on a tumor evaluation (either CT scan, physical evaluation or ultrasonography) performed less than 2 weeks before screening visit
* Requiring a treatment with Ipilimumab and PD1 inhibitor (Nivolumab) and having no contraindication to these drugs nor to their excipients
* Patients unexposed to ipilimumab and anti PD1 or anti PDL1 except if they have received it in the adjuvant setting (if the last dose of Ipilimumab® or anti PD1 or anti PDL1 was received at least 6 months before randomization).
* Negative pregnancy test (serum)
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab, ipilimumab and 6 months after the last dose of study treatment (ie, 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo approximately five half-lives)
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab, ipilimumab and 7 months after the last dose of study treatment {i.e., 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five half-lives.}
* Hemoglobin ≥9 g/dL
* Platelets ≥ 100000mm3
* Neutrophils ≥ 1500/mm3
* Creatinine Clearance ≥ 50mL/mn
* AST ≤ 3N
* ALT ≤ 3N
* Total bilirubin ≤ 1.5N (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Alkaline phosphatase ≤ 3N
* INR < 1.5
* Prothrombin ≥ 70%
* TCA < 1.2
* No Hepatocellular insufficiency

Exclusion Criteria:

* Pregnant or breastfeeding women
* Antibiotics in the last two weeks prior to the FMT
* Inability to retain enemas
* Expected to require any other form of systemic or localized anti-neoplastic therapy while on study
* Active infection requiring systemic therapy.
* Active, known or suspected autoimmune disease.
* No health insurance,
* Patients already included in a clinical research other than an observational study (e.g: registry, cohort).
* Patient on AME (state medical aid) (unless exemption from affiliation)
* Patients guardianship/legal protection/curatorship
* Contraindication to fecal transplantation
* Known hypersensitivity to Normacol or Moviprep® or equivalent patent medicines enema or one of their components.
* Fluid-electrolyte disorders with sodium retention (heart failure, hyperaldosteronism, drug-induced edema)
* Recent acute coronary syndrome or unstable ischemic heart disease
* Congestive heart failure ≥ Class III or IV as defined by New York Heart Association
* Hypersensitivity to the active substances or to any of the excipients: Aspartame (E951), Acesulfame, potassium (E950), lemon flavor (maltodextrin, citral, lemon essential oil, lime essential oil, xanthan gum, vitamin E)
* Gastrointestinal obstruction or perforation
* Gastric emptying disorders (gastroparesis),
* Ileus,
* Phenylketonuria (due to the presence of aspartame),
* Deficiency in glucose-6-phosphate dehydrogenase (due to the presence of ascorbate),
* Toxic megacolon, in severe forms of inflammation of the intestinal tract, including Crohn's disease and ulcerative colitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
To assess whether the safety of a 23-week treatment with MaaT013, combined with ipilimumab+nivolumab, is different from that of ipilimumab+nivolumab+placebo in patients with melanoma naïve to Ipilimumab and anti-PD1 | During the 27 weeks of the trial.
  Safety will be measured by the occurrence of treatment-related adverse events of Grade 3, grade 4 and grade 5, as graded by the CTCAE v 5.0, during the 27 weeks of the trial

SECONDARY OUTCOMES:
To assess whether a 23-week treatment with MaaT013, combined with Ipilimumab and Nivolumab, is more efficient than Ipilimumab and Nivolumab + placebo in patients with melanoma naïve to Ipilimumab and anti PD1. | During the 27 weeks of the trial.
  Efficacy will be assessed by the best overall response rate, between baseline and week 27, without confirmation of partial or complete response rated by Response Evaluation Criteria in Solid Tumors (RECIST v1.1.; 19) in the experimental and control arms.
To assess changes in the tumor microenvironment in patients who have received MaaT013 and placebo ; | During the 27 weeks of the trial.
  Changes in the tumor micro environment (TME) pre and post MaaT013 or placebo
Changes in plasma levels of proteins or metabolites that play a role in immune activity against cancer and/or are associated with gut microbiome composition, pre and post MaaT013 or placebo | During the 27 weeks of the trial.
  Changes in plasma levels of proteins or metabolites that play a role in immune activity against cancer and/or are associated with gut microbiome composition, pre and post MaaT013 or placebo : IL-6, IL-8, MCP1, IL-1β, TNF α, sCD25, sCTLA-4, sPD-L1, short chain fatty acids (SCFA), all in micromol/L
Changes in signatures of peripheral blood T or immune cells cell. T cell or other immune cells will be sorted and transcriptomic analysis will be performed to determine changes induce by MaaT013 or placebo treatment. | During the 27 weeks of the trial.
  Changes in peripheral blood immune cell subpopulations pre and post MaaT013 or placebo
To assess the evolution of gut microbial members and metabolites; | During the baseline and 9 weeks of the trial.
  Changes in gut microbiome and metabolites pre and post MaaT013 or placebo and in patients who met the inclusion criteria, received Ipilimumab+Nivolumab, agreed to have stool microbiome analyses at baseline and week 9, but did not receive MaaT013 or placebo.
To assess, on an open basis, the efficacy and safety of MaaT013 combined with Nivolumab in a subset of patients who failed to respond to placebo | During the 51 weeks of the trial.
  Best response rate, either complete or partial, rated by RECIST and iRECIST in patients with disease progression who received placebo and subsequently, MaaT013, in an open-label basis
To assess progression-free survival at week 15, 27, 51 | During the 15, 27 and 51 weeks of the trial.
  Progression-free survival rated by RECIST and iRECIST at week 15, 27 and 51
To assess response (either partial or complete), stable disease and progression at week 15, 27, 51 | During the 15, 27 and 51 weeks of the trial.
To assess overall survival at week 15, 27, 51. | During the 15, 27 and 51 weeks of the trial.
  Time point assessment of response (either partial or complete), stable disease and progression at week 15, 27 and 51
To assess best overall response rate, either complete or partial, with or without confirmation of response, rated by iRECIST v1.1 and PET scan at weeks 15, 27 and 51, using EORTC criteria | During the 15, 27 and 51 weeks of the trial.
  Best overall response rate, either complete or partial, with or without confirmation of response, rated by iRECIST v1.1. (20) and PET scan at weeks 15, 27 and 51, using EORTC criteria
Best overall response rate, with confirmation of response, rated by RECIST (19) | During the 27 weeks of the trial.
  Best overall response rate, without confirmation of response between baseline and week 27, rated by RECIST (19)
To assess disease control rate (complete or partial response or stable disease) | During the 15, 27 and 51 weeks of the trial.
  Disease control rate (complete or partial response or stable disease) rated by RECIST and iRECIST
To assess pseudo progression rate | During the 15, 27 and 51 weeks of the trial.
  Pseudo progression rate evaluated by iRECIST
The description of favorable gut microbiome will be based upon analyses performed in patients of the placebo arm, | During the 27 weeks of the trial.
  This is why patients who met the inclusion criteria, received Ipilimumab+Nivolumab, who consented to have gut microbiome analyses at baseline and week 9, but were not included in the randomized trial, will be followed until week 27.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Ambroise Paré, Boulogne-Billancourt, Boulogne-Billancourt
  - Hôpital Lille, Lille, Lille
  - Hôpital Nantes Hôtel Dieu, Nantes, Nantes
  - Hôpital Saint Louis, Paris, Paris
  - Hôpital Gustave Roussy, Villejuif, Villejuif